CLINICAL TRIAL: NCT00940524
Title: Phase I Study of Induction Therapy With Cytarabine, High-Dose Mitoxantrone and Dasatinib for Patients With Philadelphia-Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia (ALL): ALL-6 Protocol
Brief Title: Induction Therapy With Cytarabine, High-Dose Mitoxantrone and Dasatinib for Patients With Philadelphia-Chromosome Positive (Ph+) Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-046
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Leukemia; Acute Lymphoblastic Leukemia
Keywords: Leukemia; ALL; ALLOPURINOL; CARMUSTINE (BCNU); CYCLOPHOSPHAMIDE (CYTOXAN); CYTARABINE (ARA-C); DACTINOMYCIN; DASATINIB; DEXAMETHASONE; DOXORUBICIN/ADRIAMYCIN; ETOPOSIDE (VP-16); MERCAPTOPURINE; METHOTREXATE; MITOXANTRONE; PEGASPERGASE; VINCRISTINE
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib; Mitoxantrone; Cytarabine; Cyclophosphamide; Aging; Etoposide; pegaspargase; Asparaginase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): A phase I study designed to determine the dose of dasatinib that can be safely administered with cytarabine and high-dose mitoxantrone in Ph+ ALL / lymphoid blast crisis of known chronic myelogenous leukemia patients.
  Interventions: Drug: Dasatinib, Mitoxantrone, Cytarabine

INTERVENTIONS:
Drug: Dasatinib, Mitoxantrone, Cytarabine — INDUCTION- Dasatinib† (dose levels 1-3) *continuously Cytarabine 3 g/m2 IV over 3 hours Mitoxantrone 80 mg/m2 IV Myeloid growth factor on day 7 until ANC > 1,000/μl x 2 days Allopurinol 300 mg BID-TID x 7 days (starting 6-12 hours prior to chemotherapy) Dexamethasone 0.1% eye drops q6h while on cytarabine (start prior to the first dose of cytarabine and continuing at least 24 hours after the last dose) IT Methotrexate 12 mg days 2 and 4
  CONSOLIDATION A-Dasatinib† (dose levels 1-3) *continuously Vincristine 2 mg IV Dexamethasone 10 mg/m2/d days 2 to 29, then taper over 10 days Sulfamethoxazole/Trimethoprim 1 DS BID three times weekly days 2 to 29, then BID daily days 30 to 45 IT Methotrexate 12 mg days 8, 15, 22 and 29
  Other Names: CONSOLIDATION B-Dasatinib† (dose levels 1-3) *continuously; Cyclophosphamide 4 g/m2 IV (age > or = 60 yrs 3 g/m2); Myeloid growth factor on day 7 until ANC > 1,000/μl x 2 days; CONSOLIDATION C-Dasatinib† (dose levels 1-3) *continuously; Cytarabine 200 mg/m2/d IVCI (continuous infusion); Etoposide 200 mg/m2/d IV; IT Methotrexate 12 mg x 2 (between days 1-7); CONSOLIDATION D-Dasatinib† (dose levels 1-3) *continuously; Pegaspargase 2,000 IU/m2 IV (preferred) or IM day 1 (Patients age > or = 60 yrs receive 1,000 IU/m2); *If Pegaspargase is unavailable, L-asparaginase should be substituted; L-asparaginase 10,000 IU/m2/d IV (preferred) or IM, three times weekly x 6 doses; (Patients age > or = 60 yrs receive 6,000 IU/m2/d IV or IM, three times weekly x 6 doses); Patients in CR will proceed to Maintenance therapy.

SUMMARY:
This research study is for people with a specific type of leukemia called Philadelphia chromosome positive acute lymphoblastic leukemia (the type the patients have). The investigators plan to give you combination of 3 drugs (dasatinib, mitoxantrone, cytarabine) for the first part of the chemotherapy (called Induction). The investigators have previously shown that the combination of mitoxantrone and cytarabine is very effective in your kind of leukemia. The purpose of this study is to establish a safe dose range of dasatinib in combination with this standard induction chemotherapy based on side effects. If possible, the trial will also give us an idea of how well this combination might work in treating your leukemia. Previous studies have shown that dasatinib can produce responses when given alone for your kind of leukemia. By using the dasatinib together with the chemotherapy, the investigators believe that we can kill even more leukemia cells than with either treatment alone. The investigators will initially treat patients with a low dose of dasatinib and monitor for side-effects. If the initial group of patients is able to tolerate this low-dose of dasatinib, then future patients will receive higher doses of dasatinib. Mitoxantrone and cytarabine chemotherapy is the standard therapy at the investigators' institution for the patient's leukemia and it is the combination of dasatinib with this chemotherapy that is new and investigational in this study.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated and treated adult patients (> or = 18 years old) with a diagnosis of:

  * Philadelphia-chromosome positive acute lymphoblastic leukemia
  * Lymphoid blast crisis of known chronic myelogenous leukemia NOTE: Patients must have evidence of a t(9;22) in leukemic cells based on chromosomal or molecular analysis.

NOTE: The diagnosis must be confirmed by the pathology department at MSKCC. NOTE: It is recognized that newly diagnosed patients may be started on therapy with cytarabine and high-dose mitoxantrone (which is the standard of care at our institution for treating adult ALL) prior to the identification of t(9;22) in leukemic cells. These patients will remain eligible for participation on study and will be evaluable for response if it is possible to start treatment with dasatinib within 30 days of receiving induction chemotherapy.

* Patients with adequate hepatic function (AST and ALT < or = 2.5 the institutional ULN, bilirubin < or = 2.0 mg/dl).
* Patients with adequate renal function (creatinine < or = 2.0 mg/dl or creatinine clearance > 50 ml/min).
* Patients with an LVEF > or = 50%.
* Karnofsky performance status > or = 20%.
* Ability to take oral medication (dasatinib must be swallowed whole).
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (sensitivity > or = 25IU HCG/L) within 72 hours prior to the start of study drug administration. Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study drug is stopped. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* concomitant Medications: Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy (discontinue St. Johns Wort at least 5 days before starting dasatinib); Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
* Signed informed consent, which indicates the investigational nature of this study, within 30 days of treatment initiation, is required.

Exclusion Criteria:

* Female patients who are pregnant or lactating. Women and men of childbearing age should use effective contraception.
* Patients with uncontrolled active infections.
* Patients who are receiving other systemic chemotherapy. Patients must have been off prior antileukemic therapy for at least 2 weeks (hydroxyurea is considered acceptable).

NOTE: Patients who had previously received combination therapy with cytarabine, high-dose mitoxantrone and dasatinib will be excluded from the trial. All other prior therapies will be allowed, including prior tyrosine kinase inhibitors usage. Prior dasatinib use will be allowed (as a single agent or in combination therapy, other than the combination therapy with cytarabine and high-dose mitoxantrone).

* Concomitant active secondary malignancy requiring treatment (other than squamous cell and basal cell carcinoma of skin).
* Concurrent medical condition which may increase the risk of toxicity, including: grade ≥ 2 pleural or pericardial effusion.
* Cardiac Symptoms; any of the following should be considered for exclusion:

  * Uncontrolled angina, congestive heart failure or MI within (6 months).
  * Diagnosed congenital long QT syndrome.
  * Any history of clinically significant ventricular arrhythmias (such as ventricular - tachycardia, ventricular fibrillation, or Torsades de pointes).
  * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec).
  * Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration.
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease).
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).

Ongoing or recent (< or = 3 months) significant gastrointestinal bleeding

* Concomitant Medications, any of the following should be considered for exclusion:

  * Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib)
  * quinidine, procainamide, disopyramide amiodarone, sotalol, ibutilide, dofetilide erythromycin, clarithromycin chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To determine the dose of dasatinib that can be safely administered with cytarabine, and high-dose mitoxantrone in patients with Ph+ ALL / lymphoid blast crisis of known chronic myelogenous leukemia. | 5 years

SECONDARY OUTCOMES:
To determine the toxicity of this combination in these patients. | 5 years
To determine Abl-mutational status at baseline and at the time of disease progression as a possible mechanism of resistance. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Renier Brentjens, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm